CLINICAL TRIAL: NCT02636842
Title: A Phase 1, Randomized, Open-label, Single Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Aripiprazole Lauroxil Following Administration to the Deltoid or Gluteal Muscle in Adults With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study of Aripiprazole Lauroxil in Subjects With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK9072-A106
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Aripiprazole Lauroxil; Aripiprazole; ALKS 9072; Alkermes
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — aripiprazole lauroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Location (Other): Deltoid or Gluteal Muscle
  Interventions: Drug: Aripiprazole Lauroxil

INTERVENTIONS:
Drug: Aripiprazole Lauroxil — Intramuscular (IM) injection, single dose
  Other Names: ARISTADA TM

SUMMARY:
The study will determine the safety, tolerability, and pharmacokinetics of aripiprazole lauroxil in adults with schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of chronic schizophrenia or schizoaffective disorder
* Has demonstrated ability to tolerate aripiprazole
* Has been on a stable antipsychotic medication regimen without any changes for at least 2 months prior to screening
* Has a body mass index (BMI) of 18.0 to 40.0 kg/m2, inclusive
* Additional criteria may apply

Exclusion Criteria:

* Is pregnant, is planning to become pregnant, or is currently breastfeeding
* Has received aripiprazole lauroxil or IM depot aripiprazole within 6 months, or other long-acting, injectable antipsychotic medication within 3 months or currently treated with clozapine
* Is a danger to himself/herself at screening or upon admission
* Has a history of or positive test result for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Has a positive urine drug screen at screening or Day 1
* Additional criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 7 days

SECONDARY OUTCOMES:
Time to Cmax (Tmax) | Up to 7 days
Area under the concentration-time curve from time zero to the last quantifiable time interval (AUCl0-last) | Up to 7 days
Area under the concentration-time curve from time zero to time t (AUC0-t) | Up to 7 days
Terminal elimination half-life (t½) | Up to 7 days
Safety will be determined by incidence of adverse events | Up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Director — Alkermes, Inc.
Locations (6):
- United States (6):
  - Alkermes Investigational Site, Cerritos, California
  - Alkermes Investigational Site, Lemon Grove, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Marlton, New Jersey
  - Alkermes Investigative Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No